CLINICAL TRIAL: NCT04583904
Title: Prospective Evaluation of Novel Diagnostics for Tuberculosis in KwaZulu-Natal, South Africa
Acronym: PROVE-TB
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Umkhuseli Innovation and Research Management (UIRM) (Unknown); University of KwaZulu (Other); PATH (Other); KwaZulu Natal Department of Health (Unknown); Salus Ltd. (Industry)
Responsible Party: Principal Investigator, Paul Drain, Associate Professor of Global Health, Medicine and Epidemiology, University of Washington
Other Study IDs: STUDY00009092; OPP1213504 (Other Grant/Funding Number: Bill & Melinda Gates Foundation)
Record Dates: First submitted 2020-09-29; First posted 2020-10-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis
Keywords: Urine-Lam; Diagnostics
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, urine, whole blood, PBMC, oral fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults - inpatient
- Adults- ambulatory
- Children

SUMMARY:
Tuberculosis (TB) infects nearly two billion people and has become the leading infectious cause of mortality worldwide, due in part to inadequate diagnostic and prognostic tests. Older diagnostic tools, such as acid-fast staining, and newer diagnostic tests, such as nucleic acid amplification, are either insensitive, expensive, or not suitable for use at the clinical point-of-care. Therefore, novel diagnostic tests are needed to diagnose active TB disease among adults, people living with HIV (PLHIV), and children in TB-endemic countries. In this project, the investigators will conduct clinical evaluation studies of emerging TB diagnostic tests among (1) hospitalized adults, (2) ambulatory adults in outpatient clinics, and (3) children <12 years suspected of having active TB disease. the investigators will also maintain a biorepository of well-characterized clinical specimens that can be used for either retrospective validation of TB diagnostic tests, establishing a reference LAM test, or to share with partners developing novel TB diagnostics, including new LAM antibodies. The project will be coordinated at the University of Washington, and conducted in partnership with clinical research partners in South Africa, including Umkhuseli Innovation and Research Management (UIRM) and the National Health Laboratory Service (NHLS). The project team is well-equipped to serve as a central clinical research site to evaluate new and emerging point-of-care TB diagnostics, particularly novel urinary LAM assays, at the on-site TB Diagnostics Research Laboratory at Edendale Hospital in KwaZulu-Natal, South Africa.

ELIGIBILITY:
Phase I

1. Eligibility for hospitalized and ambulatory adults:

* ≥16 years old
* Positive Xpert MTB/RIF Ultra test (TB-positive cohort) or no suspicion of clinical TB (TB-negative cohort)
* Have a documented HIV test result or agrees to test for HIV
* Have NOT received IPT within prior 3 months
* Have NOT received anti-TB treatment for more than 24 hours
* Willing/able to provide written informed consent

Phase II:

1. Eligibility for hospitalized adults:

   * ≥16 years old
   * Admitted to inpatient medical ward <72 hours
   * Have a documented positive HIV test
   * Have NOT received IPT within prior 3 months
   * Have NOT received anti-TB treatment for more than 24 hours
   * Willing/able to provide written informed consent

   Study population description:
2. Eligibility for Xpert+ adults (hospitalized and attending outpatient clinics)

   * ≥16 years old
   * Have a documented HIV test result or agrees to test for HIV
   * Positive Xpert MDR/RIF Ultra test documented.
   * Have NOT received anti-TB treatment for more than 24 hours
   * Willing/able to provide written informed consent

     3) Eligibility for children
   * children <12 years of age
   * suspected of having active TB disease by clinical team
   * Have a documented HIV test result or agrees to test for HIV
   * Have not had IPT within 3 months
   * Have not received anti-TB treatment for more than 24 hours within the prior 5 days
   * Parent or guardian is willing/able to provide written informed consent

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study may enroll 3 different types of patient cohorts, including (1) hospitalized adults (≥16 years old), (2) ambulatory adults (≥16 years old) in outpatient clinics, and (3) children <12 years suspected of having active TB disease.
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants Classified with TB Case Definition | Baseline
  TB positive: A person with a positive Xpert MTB/RIF test or TB culture on any bodily fluid specimen that was obtained/tested within 5 days of enrollment.
  Probable TB: A person with compatible symptoms, signs, histopathological specimens and imaging for TB, but without a positive TB culture or Xpert test on any specimen; empirically initiated on TB treatment.
  TB negative: A person with a primary hospital diagnosis other than TB, who has no clinical suspicion for TB, and no diagnostic TB testing ordered by the treating team.
  TB negative (TB excluded): A person with all reference microbiological testing for TB returning negative, including negative Xpert, negative TB culture, other investigations for TB negative (e.g. histopathology, imaging) and either clinical improvement in the absence of anti-TB therapy or alternate diagnosis determined. In addition, no incident TB diagnosis made (including empiric anti-TB treatment initiation) within the 2 months following enrollment.

SECONDARY OUTCOMES:
Number of Participants with TB Treatment Outcome | 2 Month, 6 Month
  * Confirmed TB: Bacteriological confirmation obtained: culture or Xpert MTB/RIF from at least one specimen.
  * Probable TB: Bacteriological confirmation not obtained AND at least 2 of the following:
  * Symptoms/signs suggestive of TB (as defined)
  * Chest radiograph or abdominal ultrasound consistent with TB
  * Close TB exposure or immunologic evidence of M. tuberculosis infection
  * Positive response to anti-TB treatment (requires documented positive clinical response on TB treatment)
  * TB negative/unlikely: Bacteriological confirmation NOT obtained AND criteria for "unconfirmed tuberculosis" NOT met.

CONTACTS AND LOCATIONS:
Overall Officials: Paul K. Drain, MD, MPH, FACP, Principal Investigator — University of Washington; Douglas Wilson, MD, Principal Investigator — University of KwaZulu
Locations (1):
- Edendale Hospital, Pietermaritzburg, South Africa

IPD SHARING:
Plan to Share IPD: Undecided